CLINICAL TRIAL: NCT04504955
Title: CorEvitas Atopic Dermatitis Registry: A Study of Post Approval Drug Safety and Effectiveness
Status: Enrolling by invitation | Type: Observational
Sponsor: CorEvitas (Network)
Responsible Party: Sponsor
Other Study IDs: CorEvitas-AD-550
Record Dates: First submitted 2020-07-30; First posted 2020-08-07 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimen collection is optional.It will consist of biospecimens (peripheral blood serum, plasma, DNA, and RNA)) for biobanking, biomarker, and other related analysis linked to registry (patient and provider reported) data and imaging
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atopic Dermatitis: Pts presenting to enrolling sites across in North America and select European countries are invited to enroll if eligible
  Interventions: Other: Observational Non-Interventional Registry

INTERVENTIONS:
Other: Observational Non-Interventional Registry — Observational Non-Interventional Registry

SUMMARY:
This prospective, non-interventional research registry is designed to study the comparative effectiveness and comparative safety of approved treatments for patients with atopic dermatitis under the care of a licensed dermatologist or qualified physician extender. Secondary objectives include analyzing the epidemiology and natural history of the disease, its comorbidities, and current treatment practices.

Condition or disease :

Atopic Dermatitis

DETAILED DESCRIPTION:
The objective of the CorEvitas Atopic Dermatitis (AD) Registry is to create a national cohort of patients with atopic dermatitis. Data collected will be used to extensively evaluate the effectiveness and safety of medications used to treat atopic dermatitis. This will be done through the standardized collection of patient-reported outcomes (PRO) and clinician-reported outcomes (ClinRO), and the prevalence and incidence of comorbidities and adverse events, medication utilization patterns, and patient productivity measures.

ELIGIBILITY:
Inclusion Criteria Has been diagnosed with AD by a dermatologist or qualified dermatology provider.

2) Is at least 18 years of age or older and has attained the legal age for consent to procedures involved in the research, under the applicable law of the jurisdiction in which the research is being conducted.

3) Willing and able to provide consent for participation in the registry. 4) Willing and able to provide Personal Information (full legal name, sex, date of birth, home address zip/postal code, and email address OR phone number at a minimum) if required based on registry location and applicable laws and regulations. 5) Has been prescribed a new Enrollment Eligible Medication. A new therapy is a medication that the subject has never taken before.

1. At the time of registry enrollment OR
2. Within 12 months prior to registry enrollment

Exclusion Criteria:

1)Is participating or planning to participate in a blinded clinical trial for an AD drug.

Follow-Up Criteria

Registry Follow-Up data collection should be done at the time of routine clinical encounters approximately every 6 months. Routine or standard of care clinical encounters may occur in between two registry visits, but the data collected in the Follow-Up forms should cover the time period since the last registry visit.

For planning purposes, each Follow-Up visit is anchored to the date of the last eligible registry visit. A Follow-Up visit is eligible for payment if 150 days have passed since the last visit submission. A Follow-Up visit is not eligible for payment if conducted less than 150 days since the last registry visits except when the EARLY Follow-Up visit Criteria are satisfied.

EARLY Follow-Up Criteria

A registry Follow-Up visit should be conducted whenever a patient is prescribed or receiving the first dose of a new Eligible Medication even if less than 150 days have passed since the last registry visit. When the EARLY Follow-Up criteria are met, the next anticipated registry visit is calculated from the date of the Early Follow-Up visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are enrolled in the Atopic Dermatitis Registry during regularly scheduled office visits clinical encounters. Selected dermatologists are invited to participate as investigators in the Registry.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2100-12 (Estimated); Study Completion 2100-12 (Estimated)

PRIMARY OUTCOMES:
AD epidemiology, presentation, natural history, management, and outcomes | Through Study completion, an average of 10years
  The major clinical outcomes include an assessment of the epidemiology of Atopic Dermatitis; to better understand the presentation, natural history, management and outcomes.

SECONDARY OUTCOMES:
Percentage of patients with history of comorbidities | at registry enrollment
Physician reported: validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) | every 6 months for 10 years
  Score: 0-4, with high score indicating widespread of atopic dermatitis
Physician reported: Nail changes due to atopic dermatitis (graduated VAS) | every 6 months for 10 years
  Scale - 0 (Clear/Normal) to 100 (Severe Abnormalities). Lower numbers are for mild abnormalities in a few nails, higher numbers are for more severe changes in many nails
Physician reported: Atopic dermatitis body surface area (BSA) | every 6 months for 10 years
Physician reported: Eczema Area and Severity Index (EASI) (calculated) | every 6 months for 10 years
  The severity of each sign will be graded on a scale of 0 to 3: (0) None, (1) Mild, (2) Moderate, (3) Severe.
Physician reported : SCORing Atopic Dermatitis index (SCORAD) (calculated) | every 6 months for 10 years
  The severity of each sign will be graded on a scale of 0 to 3: (0) None, (1) Mild, (2) Moderate, (3) Severe. For the Overall Score [SCORAD], select a lesion that that is representative of the body and score using the same severity scale
Patient reported: Patient global assessments of disease control and severity | every 6 months for 10 years
  This determines the progression & severity of the disease
Patient reported: Patient Oriented Eczema Measure (POEM) | every 6 months for 10 years
Patient reported: Peak pruritus (itch) NRS | every 6 months for 10 years
Patient reported: Skin pain NRS | every 6 months for 10 years
Patient reported: Fatigue NRS | every 6 months for 10 years
Patient reported: Dermatology Life Quality Index (DLQI) | every 6 months for 10 years
Patient reported: Work Productivity and Activity Impairment (WPAI) | every 6 months for 10 years
Patient reported: Atopic dermatitis control tool (ADCT) | every 6 months for 10 years
Patient reported: Itch triggers (PROMIS) | every 6 months for 10 years
Patient reported: Sleeplessness and average pruritus (itch) NRS (SCORAD) | 6 months for 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- CorEvitas, LLC, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No